CLINICAL TRIAL: NCT01111019
Title: Efficacy and Safety Evaluation of Recombinant Human Growth Hormone (r-hGH), Saizen®, on a Population of Children With Hypochondroplasia, Treated Over a Period of 3 Years or 5 Years if Applicable, in Comparison With a Historic Cohort of Non-treated Children With Hypochondroplasia
Brief Title: Efficacy and Safety Evaluation of Recombinant Human Growth Hormone (r-hGH), Saizen®, on a Population of Children With Hypochondroplasia, Treated at Least 3 Years or Until Near Final Height, When Applicable, in Comparison With a Historic Cohort of Non-treated Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono S.A.S, France (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMP 26545 (EMR701048-506)
Record Dates: First submitted 2010-04-23; First posted 2010-04-27 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-10

CONDITIONS: Hypochondroplasia
Keywords: Hypochondroplasia; Skeletal dysplasia; Growth; Growth Hormone; Recombinant-human Growth Hormone
MeSH Terms: conditions — Hypochondroplasia; Mucopolysaccharidosis IV | interventions — Growth Hormone; Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- r-hGH (Saizen®) (Experimental)
  Interventions: Drug: Recombinant human growth hormone (r-hGH)

INTERVENTIONS:
Drug: Recombinant human growth hormone (r-hGH) — Subjects will receive a single subcutaneous injection of recombinant human growth hormone (r-hGH) equivalent to a dose of 0.057 milligram per kilogram per day (mg/kg/day). The dose will be subsequently adjusted during the trial and subjects will be treated for at least 3 years or until near final height is reached.
  Other Names: Saizen®, Somatropin

SUMMARY:
This study is conducted to describe the efficacy and safety of recombinant human growth hormone (r-hGH) treatment Saizen® on children with hypochondroplasia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female children with hypochondroplasia defined by a disproportional short limb height and a X-ray evidence of shortening of the long bones and failure of increase in the interpedicular distance between lumbar vertebrae L1 and L5
* Result of genetic analysis for mutation of gene FGFR3 already known or ongoing analysis at the beginning of the study
* Chronological age greater than or equal to 3 years
* Height for chronological age less than or equal to - 2 SDS
* Bone age less than or equal to 11 years for girls and 13 years for boys
* A written informed consent at the beginning of the pre-treatment period must be obtained from the parent(s)/legal guardian(s). Children able to understand the trial should personally sign and date the written informed consent

Additional inclusion criteria for each study prolongation:

* Bone age at Month 36 or Month 60 is compatible with treatment prolongation according to investigator opinion
* Subject is still under r-hGH treatment with Saizen® at Month 36 or Month 60
* Height gain greater than or equal to + 1 SDS after the 2 first years of treatment for treatment prolongation at Month 36 and growth velocity greater than or equal to 5 centimeter (cm) per year, with bone age less than 14 years for females or less than 16 years for males for treatment prolongation at Month 60
* According to investigator opinion, gene mutations of the subjects are not in connection with observed side effects during the 3 or 5 first years of treatment
* An updated written informed consent must be obtained from the parent(s)/legal guardian(s) before the start of each study prolongation. Children able to understand the trial should personally sign and date the written informed consent

Exclusion Criteria:

* Turner's Syndrome in girls
* Active malignant neoplastic disease
* Severe congenital malformations
* Proliferative or preproliferative diabetic retinopathy
* Evidence of any progression or recurrence of an underlying intra-cranial space occupying lesion
* Severe psychomotor retardation
* Diabetes mellitus or history of significant glucose intolerance as defined by a fasting blood glucose greater than 6.4 millimole per liter (mmol/L)
* Known renal insufficiency as defined by serum creatinine level 1.0 milligram per deciliter (mg/dL) (88 micromole per liter [mcmol/L])
* Known hepatic disease as defined by elevated liver enzymes or total bilirubin (* 2 Normal)
* Current congestive heart failure, untreated hypertension, serious chronic edema of any cause
* Chronic infectious disease
* History of intracranial hypertension with papilledema
* Previous or ongoing treatment with sex steroid therapy such as estrogens or testosterone
* Previous or ongoing treatment with any therapy that may directly influence growth, including Growth Hormone (GH), Growth Hormone Releasing Hormone (GHRH) and long duration corticosteroids therapy
* Known hypersensitivity to somatropin or any of the excipients
* Epiphyseal fusion
* Participation to any clinical study within the 30 days preceding study entry
* Pregnant females

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-03-21 (Actual); Primary Completion 2017-01-17 (Actual); Study Completion 2017-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Endocrinologie Pédiatrique - centre des maladies rares de la croissance -Hôpital Necker Enfants Malades, Paris, France

REFERENCES:
- [Derived] Pinto G, Cormier-Daire V, Le Merrer M, Samara-Boustani D, Baujat G, Fresneau L, Viaud M, Souberbielle JC, Pineau JC, Polak M. Efficacy and safety of growth hormone treatment in children with hypochondroplasia: comparison with an historical cohort. Horm Res Paediatr. 2014;82(6):355-63. doi: 10.1159/000364807. Epub 2014 Oct 15. PMID 25323764

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between March 21, 2006 and January 17, 2017.
Groups:
- r-hGH (Saizen®): Subjects received a single subcutaneous injection of recombinant human growth hormone (r-hGH) equivalent to dose of 0.057 milligram per kilogram per day (mg/kg/day). The dose was subsequently reduced to 0.035 mg/kg/day for subjects, who continued treatment after 31 January 2011. Subjects were treated for at least 3 years or until near final height was reached.
Period: Overall Study
Arm/Group | r-hGH (Saizen®)
Started | 19
Completed | 16
Not Completed | 3
Not completed — Withdrew Prematurely | 2
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: Intention to Treat (ITT) population included all subjects who received at least one dose of treatment with at least an efficacy assessment available during the treatment period.
Arm/Group | r-hGH (Saizen®)
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.0 (3.12)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 11
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Height-Standard Deviation Score (H-SDS) of Recombinant Human Growth Hormone (r-hGH) Treated Subjects at Year 3
Description: Height was calculated in standardized units expressed as the standard deviation score (SDS), where SDS = (x - m)/sigma, in which x represents the height variable measured by sex and age, and m and sigma are the statistical parameters (mean and standard deviation) for the Sempe reference population. The reference population was the historical cohort consisting of non-treated subjects with Hypochondroplasia (HCH). SDS indicated how many standard deviations higher (in case of positive SDS) or lower (in case of negative SDS) a participant's value was relative to the mean of the reference population. The scores were centered around zero. Negative score indicated smaller height for the respective age/gender.
Time Frame: Baseline (Month 0), Year 3
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Standard Deviation Score (SDS)
Arm/Group | r-hGH (Saizen®)
Number analyzed (Participants) | 19
Standard Deviation Score (SDS) | 1.39 (0.9)

2. Primary Outcome: Height-Standard Deviation Score (H-SDS) of Recombinant Human Growth Hormone (r-hGH) Treated Subjects at Year 4
Description: as for outcome 1
Time Frame: Year 4
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Standard Deviation Score (SDS)
Arm/Group | r-hGH (Saizen®)
Number analyzed (Participants) | 19
Standard Deviation Score (SDS) | 25.6 (3.5)

3. Secondary Outcome: Height-Standard Deviation Score (H-SDS) of Recombinant Human Growth Hormone (r-hGH) Treated Subjects
Description: Height was calculated in standardized units expressed as the standard deviation score (SDS), where SDS = (x - m)/sigma, in which x represents the height variable measured by sex and age, and m and sigma are the statistical parameters (mean and standard deviation) for the Sempe reference population. The reference population was the historical cohort consisting of non-treated subjects with Hypochondroplasia (HCH). Data was reported by gender. Male subjects were analyzed till 9.5 years and female subjects were analyzed till 8.5 years. SDS indicated how many standard deviations higher (in case of positive SDS) or lower (in case of negative SDS) a participant's value was relative to the mean of the reference population. The scores were centered around zero. Negative score indicated smaller height for the respective age/gender.
Time Frame: Year 1, 2, 3, 4, 5, 6, 7, 8 (both male and female); 8.5 (only for female), 9 (only for male) and 9.5 (only for male)
Population: Intention to Treat (ITT) population included all subjects who received at least one dose of treatment with at least an efficacy assessment available during the treatment period. Here "Number analyzed" signifies those subjects who were evaluable for this outcome measure for specified category.
Measure: Median (Full Range); unit: Standard Deviation Score (SDS)
Arm/Group | r-hGH (Saizen®)
Number analyzed (Participants) | 19
Standard Deviation Score (SDS)
  Male: Year 1: number analyzed (Participants) | 8
  Male: Year 1 | -1.82 [-3.4 to -1.4]
  Male: Year 2: number analyzed (Participants) | 8
  Male: Year 2 | -1.51 [-3.4 to -1.1]
  Male: Year 3: number analyzed (Participants) | 8
  Male: Year 3 | -1.30 [-3.7 to -1.0]
  Male: Year 4: number analyzed (Participants) | 4
  Male: Year 4 | -1.49 [-3.7 to -1.0]
  Male: Year 5: number analyzed (Participants) | 4
  Male: Year 5 | -1.51 [-3.5 to -1.0]
  Male: Year 6: number analyzed (Participants) | 2
  Male: Year 6 | -2.88 [-3.8 to -2.0]
  Male: Year 7: number analyzed (Participants) | 1
  Male: Year 7 | -3.9 [-3.9 to -3.9]
  Male: Year 8: number analyzed (Participants) | 1
  Male: Year 8 | -3.90 [-3.9 to -3.9]
  Male: Year 9: number analyzed (Participants) | 1
  Male: Year 9 | -5.0 [-5.0 to -5.0]
  Male: Year 9.5: number analyzed (Participants) | 1
  Male: Year 9.5 | -5.6 [-5.6 to -5.6]
  Female: Year 1: number analyzed (Participants) | 11
  Female: Year 1 | -2.69 [-5.3 to -0.6]
  Female: Year 2: number analyzed (Participants) | 11
  Female: Year 2 | -2.52 [-5.8 to -0.7]
  Female: Year 3: number analyzed (Participants) | 11
  Female: Year 3 | -2.61 [-6.0 to -0.6]
  Female: Year 4: number analyzed (Participants) | 4
  Female: Year 4 | -1.09 [-1.5 to -0.9]
  Female: Year 5: number analyzed (Participants) | 3
  Female: Year 5 | -1.63 [-1.9 to -1.4]
  Female: Year 6: number analyzed (Participants) | 2
  Female: Year 6 | -2.51 [-3.4 to -1.6]
  Female: Year 7: number analyzed (Participants) | 2
  Female: Year 7 | -2.74 [-3.7 to -1.8]
  Female: Year 8: number analyzed (Participants) | 1
  Female: Year 8 | -2.8 [-2.8 to -2.8]
  Female: Year 8.5: number analyzed (Participants) | 1
  Female: Year 8.5 | -3.1 [-3.1 to -3.1]

4. Secondary Outcome: Change From Baseline in Height of Recombinant Human Growth Hormone (r-hGH) Treated Subjects With Hypochondroplasia (HCH) up to 9.5 Years
Description: Body proportion was measured in terms of height. Data was reported by gender. Male subjects were analyzed till 9.5 years and female subjects were analyzed till 8.5 years.
Time Frame: Baseline (Month 0), Year 1, 2, 3, 4, 5, 6, 7, 8 (both male and female); 8.5 (only for female), 9 (only for male) and 9.5 (only for male)
Population: Intention to Treat (ITT) population included all subjects who received at least one dose of treatment with at least an efficacy assessment available during the treatment period. Here "Number Analyzed" signifies those subjects who were evaluable for the specified category.
Measure: Mean (Standard Deviation); unit: Centimeter (cm)
Arm/Group | r-hGH (Saizen®)
Number analyzed (Participants) | 19
Centimeter (cm)
  Male: Year 1: number analyzed (Participants) | 8
  Male: Year 1 | 8.10 (1.867)
  Male: Year 2: number analyzed (Participants) | 8
  Male: Year 2 | 14.59 (2.527)
  Male: Year 3: number analyzed (Participants) | 8
  Male: Year 3 | 20.00 (3.398)
  Male: Year 4: number analyzed (Participants) | 4
  Male: Year 4 | 23.74 (4.136)
  Male: Year 5: number analyzed (Participants) | 4
  Male: Year 5 | 29.06 (4.809)
  Male: Year 6: number analyzed (Participants) | 2
  Male: Year 6 | 31.35 (8.556)
  Male: Year 7: number analyzed (Participants) | 1
  Male: Year 7 | 28.40 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Male: Year 8: number analyzed (Participants) | 1
  Male: Year 8 | 34.73 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Male: Year 9: number analyzed (Participants) | 1
  Male: Year 9 | 37.98 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Male: Year 9.5: number analyzed (Participants) | 1
  Male: Year 9.5 | 38.37 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Female: Year 1: number analyzed (Participants) | 11
  Female: Year 1 | 7.72 (1.642)
  Female: Year 2: number analyzed (Participants) | 11
  Female: Year 2 | 13.76 (3.505)
  Female: Year 3: number analyzed (Participants) | 11
  Female: Year 3 | 17.95 (5.189)
  Female: Year 4: number analyzed (Participants) | 4
  Female: Year 4 | 26.96 (2.394)
  Female: Year 5: number analyzed (Participants) | 3
  Female: Year 5 | 30.08 (3.791)
  Female: Year 6: number analyzed (Participants) | 2
  Female: Year 6 | 32.50 (0.566)
  Female: Year 7: number analyzed (Participants) | 2
  Female: Year 7 | 36.92 (0.024)
  Female: Year 8: number analyzed (Participants) | 1
  Female: Year 8 | 39.47 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Female: Year 8.5: number analyzed (Participants) | 1
  Female: Year 8.5 | 40.87 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.

5. Secondary Outcome: Change From Baseline in Upper Segment (Superior) of Recombinant Human Growth Hormone (r-hGH) Treated Subjects With Hypochondroplasia (HCH) up to 9.5 Years
Description: Body proportion was measured in terms of upper segment for standing and sitting position. Data was reported by gender. Male subjects were analyzed till 9.5 years and female subjects were analyzed till 8.5 years.
Time Frame: as for outcome 4
Population: ITT population. Here "Number analyzed" signifies those subjects who were evaluable for this outcome measure for specified category. Number Analyzed was "0" at certain time points because there was no data collected at the specified time points.
Measure: Mean (Standard Deviation); unit: Centimeter (cm)
Arm/Group | r-hGH (Saizen®)
Number analyzed (Participants) | 19
Centimeter (cm)
  Male: Year 1: number analyzed (Participants) | 8
  Male: Year 1 | 3.80 (1.656)
  Male: Year 2: number analyzed (Participants) | 7
  Male: Year 2 | 7.96 (4.172)
  Male: Year 3: number analyzed (Participants) | 8
  Male: Year 3 | 8.93 (9.504)
  Male: Year 4: number analyzed (Participants) | 1
  Male: Year 4 | 16.50 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Male: Year 5: number analyzed (Participants) | 4
  Male: Year 5 | 16.98 (2.161)
  Male: Year 6: number analyzed (Participants) | 2
  Male: Year 6 | 17.05 (6.576)
  Male: Year 7: number analyzed (Participants) | 0
  Male: Year 8: number analyzed (Participants) | 0
  Male: Year 9: number analyzed (Participants) | 1
  Male: Year 9 | 18.70 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Male: Year 9.5: number analyzed (Participants) | 1
  Male: Year 9.5 | 27.80 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Female: Year 1: number analyzed (Participants) | 10
  Female: Year 1 | 4.19 (0.909)
  Female: Year 2: number analyzed (Participants) | 11
  Female: Year 2 | 9.21 (2.450)
  Female: Year 3: number analyzed (Participants) | 11
  Female: Year 3 | 13.41 (1.978)
  Female: Year 4: number analyzed (Participants) | 2
  Female: Year 4 | 15.70 (2.546)
  Female: Year 5: number analyzed (Participants) | 3
  Female: Year 5 | 15.20 (0.849)
  Female: Year 6: number analyzed (Participants) | 2
  Female: Year 6 | 18.35 (0.354)
  Female: Year 7: number analyzed (Participants) | 2
  Female: Year 7 | 21.90 (0.707)
  Female: Year 8: number analyzed (Participants) | 1
  Female: Year 8 | 24.40 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Female: Year 8.5: number analyzed (Participants) | 0

6. Secondary Outcome: Change From Baseline in Weight of Recombinant Human Growth Hormone (r-hGH) Treated Subjects With Hypochondroplasia (HCH) up to 9.5 Years
Description: The body weight was measured on a certified and calibrated hospital scale. Data was reported by gender. Male subjects were analyzed till 9.5 years and female subjects were analyzed till 8.5 years.
Time Frame: as for outcome 4
Population: ITT population. Here "Number analyzed" signifies those subjects who were evaluable for this outcome measure for specified category.
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | r-hGH (Saizen®)
Number analyzed (Participants) | 19
Kilogram (kg)
  Male: Year 1: number analyzed (Participants) | 8
  Male: Year 1 | 4.58 (2.715)
  Male: Year 2: number analyzed (Participants) | 8
  Male: Year 2 | 9.95 (4.577)
  Male: Year 3: number analyzed (Participants) | 8
  Male: Year 3 | 15.18 (6.259)
  Male: Year 4: number analyzed (Participants) | 4
  Male: Year 4 | 14.25 (3.948)
  Male: Year 5: number analyzed (Participants) | 4
  Male: Year 5 | 20.00 (7.024)
  Male: Year 6: number analyzed (Participants) | 2
  Male: Year 6 | 25.00 (11.314)
  Male: Year 7: number analyzed (Participants) | 1
  Male: Year 7 | 19.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Male: Year 8: number analyzed (Participants) | 1
  Male: Year 8 | 23.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Male: Year 9: number analyzed (Participants) | 1
  Male: Year 9 | 28.90 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Male: Year 9.5: number analyzed (Participants) | 1
  Male: Year 9.5 | 31.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Female: Year 1: number analyzed (Participants) | 11
  Female: Year 1 | 4.72 (1.537)
  Female: Year 2: number analyzed (Participants) | 11
  Female: Year 2 | 9.85 (3.946)
  Female: Year 3: number analyzed (Participants) | 11
  Female: Year 3 | 14.37 (4.905)
  Female: Year 4: number analyzed (Participants) | 4
  Female: Year 4 | 14.70 (5.510)
  Female: Year 5: number analyzed (Participants) | 3
  Female: Year 5 | 14.93 (3.101)
  Female: Year 6: number analyzed (Participants) | 2
  Female: Year 6 | 21.25 (1.061)
  Female: Year 7: number analyzed (Participants) | 2
  Female: Year 7 | 26.25 (1.061)
  Female: Year 8: number analyzed (Participants) | 1
  Female: Year 8 | 35.20 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Female: Year 8.5: number analyzed (Participants) | 1
  Female: Year 8.5 | 38.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.

7. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) of Recombinant Human Growth Hormone (r-hGH) Treated Subjects With Hypochondroplasia (HCH) up to 9.5 Years
Description: Body proportion measured as BMI. It was calculated according to the formula BMI = Weight (kilogram)/Height square (meter square). Data was reported by gender. Male subjects were analyzed till 9.5 years and female subjects were analyzed till 8.5 years.
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Kilogram per meter square (kg/m^2)
Arm/Group | r-hGH (Saizen®)
Number analyzed (Participants) | 19
Kilogram per meter square (kg/m^2)
  Male: Year 1: number analyzed (Participants) | 8
  Male: Year 1 | 0.43 (0.579)
  Male: Year 2: number analyzed (Participants) | 8
  Male: Year 2 | 1.56 (0.968)
  Male: Year 3: number analyzed (Participants) | 8
  Male: Year 3 | 2.71 (1.302)
  Male: Year 4: number analyzed (Participants) | 4
  Male: Year 4 | 2.21 (1.147)
  Male: Year 5: number analyzed (Participants) | 4
  Male: Year 5 | 3.60 (2.240)
  Male: Year 6: number analyzed (Participants) | 2
  Male: Year 6 | 5.02 (1.039)
  Male: Year 7: number analyzed (Participants) | 1
  Male: Year 7 | 4.43 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Male: Year 8: number analyzed (Participants) | 1
  Male: Year 8 | 4.57 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Male: Year 9: number analyzed (Participants) | 1
  Male: Year 9 | 6.63 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Male: Year 9.5: number analyzed (Participants) | 1
  Male: Year 9.5 | 7.60 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Female: Year 1: number analyzed (Participants) | 11
  Female: Year 1 | 0.85 (1.112)
  Female: Year 2: number analyzed (Participants) | 11
  Female: Year 2 | 2.12 (1.978)
  Female: Year 3: number analyzed (Participants) | 11
  Female: Year 3 | 3.49 (2.341)
  Female: Year 4: number analyzed (Participants) | 4
  Female: Year 4 | 2.12 (1.778)
  Female: Year 5: number analyzed (Participants) | 3
  Female: Year 5 | 2.36 (2.207)
  Female: Year 6: number analyzed (Participants) | 2
  Female: Year 6 | 4.90 (0.634)
  Female: Year 7: number analyzed (Participants) | 2
  Female: Year 7 | 6.19 (0.408)
  Female: Year 8: number analyzed (Participants) | 1
  Female: Year 8 | 9.83 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Female: Year 8.5: number analyzed (Participants) | 1
  Female: Year 8.5 | 10.71 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.

8. Secondary Outcome: Change From Baseline in Bone Mineral Density (BMD) of Recombinant Human Growth Hormone (r-hGH) Treated Subjects With Hypochondroplasia (HCH) up to 9 Years
Description: Body composition measured as BMD. It was examined at the lumbar spine (L1-L4) and determined annually by dual-energy X-ray absorptiometry. Data was reported by gender. Male subjects were analyzed till 9 years and female subjects were analyzed till 8 years.
Time Frame: Baseline (Month 0), Year 1, 2, 3, 4, 5, 6, 7, 8 (both male and female); 9 (only for male)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Gram per square centimeter (g/cm^2)
Arm/Group | r-hGH (Saizen®)
Number analyzed (Participants) | 19
Gram per square centimeter (g/cm^2)
  Male: Year 1: number analyzed (Participants) | 8
  Male: Year 1 | 0.05 (0.050)
  Male: Year 2: number analyzed (Participants) | 8
  Male: Year 2 | 0.11 (0.063)
  Male: Year 3: number analyzed (Participants) | 8
  Male: Year 3 | 0.14 (0.059)
  Male: Year 4: number analyzed (Participants) | 4
  Male: Year 4 | 0.11 (0.054)
  Male: Year 5: number analyzed (Participants) | 4
  Male: Year 5 | 0.15 (0.064)
  Male: Year 6: number analyzed (Participants) | 2
  Male: Year 6 | 0.18 (0.182)
  Male: Year 7: number analyzed (Participants) | 0
  Male: Year 8: number analyzed (Participants) | 1
  Male: Year 8 | 0.06 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Male: Year 9: number analyzed (Participants) | 1
  Male: Year 9 | 0.12 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Female: Year 1: number analyzed (Participants) | 11
  Female: Year 1 | 0.05 (0.042)
  Female: Year 2: number analyzed (Participants) | 10
  Female: Year 2 | 0.09 (0.053)
  Female: Year 3: number analyzed (Participants) | 11
  Female: Year 3 | 0.15 (0.089)
  Female: Year 4: number analyzed (Participants) | 2
  Female: Year 4 | 0.22 (0.104)
  Female: Year 5: number analyzed (Participants) | 3
  Female: Year 5 | 0.17 (0.006)
  Female: Year 6: number analyzed (Participants) | 2
  Female: Year 6 | 0.19 (0.004)
  Female: Year 7: number analyzed (Participants) | 2
  Female: Year 7 | 0.26 (0.028)
  Female: Year 8: number analyzed (Participants) | 1
  Female: Year 8 | 0.40 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.

9. Secondary Outcome: Change From Baseline in Percent Body Fat Mass of Recombinant Human Growth Hormone (r-hGH) Treated Subjects With Hypochondroplasia (HCH) up to 9 Years
Description: Body composition measured as percentage of body fat mass. It was measured by Dual X-ray absorptiometry. Data was reported by gender. Male subjects were analyzed till 9 years and female subjects were analyzed till 8 years.
Time Frame: Baseline (Month 0), Year 1, 2, 3, 4, 5, 6, 7, 8 (both male and female); 9 (only for male)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage (%) of body fat mass
Arm/Group | r-hGH (Saizen®)
Number analyzed (Participants) | 19
Percentage (%) of body fat mass
  Male: Year 1: number analyzed (Participants) | 8
  Male: Year 1 | -4.54 (2.049)
  Male: Year 2: number analyzed (Participants) | 8
  Male: Year 2 | -4.49 (3.007)
  Male: Year 3: number analyzed (Participants) | 8
  Male: Year 3 | -2.80 (3.967)
  Male: Year 4: number analyzed (Participants) | 3
  Male: Year 4 | -3.40 (4.493)
  Male: Year 5: number analyzed (Participants) | 4
  Male: Year 5 | -2.33 (5.708)
  Male: Year 6: number analyzed (Participants) | 2
  Male: Year 6 | -0.65 (11.384)
  Male: Year 7: number analyzed (Participants) | 0
  Male: Year 8: number analyzed (Participants) | 1
  Male: Year 8 | 5.70 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Male: Year 9: number analyzed (Participants) | 1
  Male: Year 9 | 1.90 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Female: Year 1: number analyzed (Participants) | 11
  Female: Year 1 | -3.50 (3.185)
  Female: Year 2: number analyzed (Participants) | 9
  Female: Year 2 | -2.27 (4.441)
  Female: Year 3: number analyzed (Participants) | 11
  Female: Year 3 | -2.74 (5.227)
  Female: Year 4: number analyzed (Participants) | 2
  Female: Year 4 | -1.40 (3.536)
  Female: Year 5: number analyzed (Participants) | 3
  Female: Year 5 | -2.50 (1.131)
  Female: Year 6: number analyzed (Participants) | 2
  Female: Year 6 | 0.05 (6.576)
  Female: Year 7: number analyzed (Participants) | 2
  Female: Year 7 | -0.50 (5.798)
  Female: Year 8: number analyzed (Participants) | 0

10. Secondary Outcome: Change From Baseline in Lean Body Mass (LBM) of Recombinant Human Growth Hormone (r-hGH) Treated Subjects With Hypochondroplasia (HCH) up to 9 Years
Description: Body composition measured as LBM. It was measured by Dual X-ray absorptiometry. Data was reported by gender. Male subjects were analyzed till 9 years and female subjects were analyzed till 8 years.
Time Frame: Baseline (Month 0), Year 1, 2, 3, 4, 5, 6, 7, 8 (both male and female); 9 (only for male)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Gram (g)
Arm/Group | r-hGH (Saizen®)
Number analyzed (Participants) | 19
Gram (g)
  Male: Year 1: number analyzed (Participants) | 8
  Male: Year 1 | 4966.46 (2670.694)
  Male: Year 2: number analyzed (Participants) | 8
  Male: Year 2 | 9134.35 (4747.742)
  Male: Year 3: number analyzed (Participants) | 8
  Male: Year 3 | 11182.24 (4126.876)
  Male: Year 4: number analyzed (Participants) | 3
  Male: Year 4 | 11599.80 (4560.877)
  Male: Year 5: number analyzed (Participants) | 4
  Male: Year 5 | 15729.38 (6102.608)
  Male: Year 6: number analyzed (Participants) | 2
  Male: Year 6 | 20667.65 (14985.50)
  Male: Year 7: number analyzed (Participants) | 0
  Male: Year 8: number analyzed (Participants) | 1
  Male: Year 8 | 15773.80 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Male: Year 9: number analyzed (Participants) | 1
  Male: Year 9 | 21713.10 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Female: Year 1: number analyzed (Participants) | 11
  Female: Year 1 | 4384.54 (1400.497)
  Female: Year 2: number analyzed (Participants) | 9
  Female: Year 2 | 6720.74 (2597.295)
  Female: Year 3: number analyzed (Participants) | 11
  Female: Year 3 | 9229.21 (2740.883)
  Female: Year 4: number analyzed (Participants) | 2
  Female: Year 4 | 11791.85 (1173.161)
  Female: Year 5: number analyzed (Participants) | 3
  Female: Year 5 | 12989.50 (83.439)
  Female: Year 6: number analyzed (Participants) | 2
  Female: Year 6 | 14860.75 (2140.483)
  Female: Year 7: number analyzed (Participants) | 2
  Female: Year 7 | 18111.60 (1239.275)
  Female: Year 8: number analyzed (Participants) | 0

11. Secondary Outcome: Growth (Height) Velocity of Recombinant Human Growth Hormone (r-hGH) Treated Subjects With Hypochondroplasia (HCH) From Year 1 up to 9.5 Years
Description: Growth velocity was calculated in terms of height velocity. It corresponded to a difference in height between current and baseline values divided by the time interval between both evaluations. Data was reported by gender. Male subjects were analyzed till 9.5 years and female subjects were analyzed till 8.5 years.
Time Frame: Year 1, 2, 3, 4, 5, 6, 7, 8 (both male and female); 8.5 (only for female), 9 (only for male) and 9.5 (only for male)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Centimeter per year (cm/year)
Arm/Group | r-hGH (Saizen®)
Number analyzed (Participants) | 19
Centimeter per year (cm/year)
  Male: Year 1: number analyzed (Participants) | 8
  Male: Year 1 | 8.21 (2.001)
  Male: Year 2: number analyzed (Participants) | 8
  Male: Year 2 | 7.26 (1.292)
  Male: Year 3: number analyzed (Participants) | 8
  Male: Year 3 | 6.55 (1.104)
  Male: Year 4: number analyzed (Participants) | 4
  Male: Year 4 | 5.88 (1.060)
  Male: Year 5: number analyzed (Participants) | 4
  Male: Year 5 | 5.77 (0.968)
  Male: Year 6: number analyzed (Participants) | 2
  Male: Year 6 | 4.98 (1.313)
  Male: Year 7: number analyzed (Participants) | 1
  Male: Year 7 | 3.92 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Male: Year 8: number analyzed (Participants) | 1
  Male: Year 8 | 4.25 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Male: Year 9: number analyzed (Participants) | 1
  Male: Year 9 | 4.11 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Male: Year 9.5: number analyzed (Participants) | 1
  Male: Year 9.5 | 3.94 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Female: Year 1: number analyzed (Participants) | 11
  Female: Year 1 | 7.53 (1.460)
  Female: Year 2: number analyzed (Participants) | 11
  Female: Year 2 | 6.64 (1.713)
  Female: Year 3: number analyzed (Participants) | 11
  Female: Year 3 | 5.86 (1.677)
  Female: Year 4: number analyzed (Participants) | 4
  Female: Year 4 | 6.57 (0.572)
  Female: Year 5: number analyzed (Participants) | 3
  Female: Year 5 | 5.89 (0.787)
  Female: Year 6: number analyzed (Participants) | 2
  Female: Year 6 | 5.13 (0.006)
  Female: Year 7: number analyzed (Participants) | 2
  Female: Year 7 | 5.06 (0.120)
  Female: Year 8: number analyzed (Participants) | 1
  Female: Year 8 | 4.69 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Female: Year 8.5: number analyzed (Participants) | 1
  Female: Year 8.5 | 4.54 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.

12. Secondary Outcome: Head Circumference Values of Recombinant Human Growth Hormone (r-hGH) Treated Subjects With Hypochondroplasia (HCH) From Year 1 up to 9.5 Years
Description: Body proportion was measured in terms of head circumference with a tape measure. Data was reported by gender. Male subjects were analyzed till 9.5 years and female subjects were analyzed till 8.5 years.
Time Frame: Year 1, 2, 3, 4, 5, 6, 7, 8 (both male and female); 8.5 (only for female), 9 (only for male) and 9.5 (only for male)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Centimeter (cm)
Arm/Group | r-hGH (Saizen®)
Number analyzed (Participants) | 19
Centimeter (cm)
  Male: Year 1: number analyzed (Participants) | 7
  Male: Year 1 | 56.11 (1.268)
  Male: Year 2: number analyzed (Participants) | 8
  Male: Year 2 | 56.53 (1.359)
  Male: Year 3: number analyzed (Participants) | 8
  Male: Year 3 | 57.38 (1.734)
  Male: Year 4: number analyzed (Participants) | 3
  Male: Year 4 | 57.33 (2.021)
  Male: Year 5: number analyzed (Participants) | 4
  Male: Year 5 | 56.88 (1.887)
  Male: Year 6: number analyzed (Participants) | 1
  Male: Year 6 | 55.50 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Male: Year 7: number analyzed (Participants) | 1
  Male: Year 7 | 57.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Male: Year 8: number analyzed (Participants) | 0
  Male: Year 9: number analyzed (Participants) | 1
  Male: Year 9 | 57.50 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Male: Year 9.5: number analyzed (Participants) | 1
  Male: Year 9.5 | 58.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Female: Year 1: number analyzed (Participants) | 9
  Female: Year 1 | 55.20 (2.379)
  Female: Year 2: number analyzed (Participants) | 8
  Female: Year 2 | 56.06 (1.841)
  Female: Year 3: number analyzed (Participants) | 11
  Female: Year 3 | 56.23 (2.453)
  Female: Year 4: number analyzed (Participants) | 1
  Female: Year 4 | 58.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Female: Year 5: number analyzed (Participants) | 3
  Female: Year 5 | 54.33 (3.512)
  Female: Year 6: number analyzed (Participants) | 2
  Female: Year 6 | 57.25 (1.768)
  Female: Year 7: number analyzed (Participants) | 2
  Female: Year 7 | 56.75 (1.061)
  Female: Year 8: number analyzed (Participants) | 1
  Female: Year 8 | 59.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Female: Year 8.5: number analyzed (Participants) | 0

13. Secondary Outcome: Osteocalcin Values of Recombinant Human Growth Hormone (r-hGH) Treated Subjects With Hypochondroplasia (HCH) From Year 1 up to 9.5 Years
Description: Osteocalcin as bone marker was analyzed with the Immunology system Elecsys. Data was reported by gender. Male subjects were analyzed till 9.5 years and female subjects were analyzed till 8.5 years.
Time Frame: Year 1, 2, 3, 4, 5, 6, 7, 8 (both male and female); 8.5 (only for female), 9 (only for male), 9.5 (only for male)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | r-hGH (Saizen®)
Number analyzed (Participants) | 19
Nanogram per milliliter (ng/mL)
  Male: Year 1: number analyzed (Participants) | 7
  Male: Year 1 | 123.06 (55.820)
  Male: Year 2: number analyzed (Participants) | 8
  Male: Year 2 | 145.00 (35.705)
  Male: Year 3: number analyzed (Participants) | 8
  Male: Year 3 | 130.13 (36.408)
  Male: Year 4: number analyzed (Participants) | 4
  Male: Year 4 | 101.00 (34.708)
  Male: Year 5: number analyzed (Participants) | 4
  Male: Year 5 | 139.25 (76.908)
  Male: Year 6: number analyzed (Participants) | 2
  Male: Year 6 | 75.50 (47.376)
  Male: Year 7: number analyzed (Participants) | 1
  Male: Year 7 | 113.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Male: Year 8: number analyzed (Participants) | 1
  Male: Year 8 | 117.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Male: Year 9: number analyzed (Participants) | 1
  Male: Year 9 | 159.80 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Male: Year 9.5: number analyzed (Participants) | 1
  Male: Year 9.5 | 131.60 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Female: Year 1: number analyzed (Participants) | 10
  Female: Year 1 | 148.00 (46.183)
  Female: Year 2: number analyzed (Participants) | 11
  Female: Year 2 | 122.82 (46.531)
  Female: Year 3: number analyzed (Participants) | 11
  Female: Year 3 | 94.73 (33.344)
  Female: Year 4: number analyzed (Participants) | 4
  Female: Year 4 | 102.00 (26.268)
  Female: Year 5: number analyzed (Participants) | 3
  Female: Year 5 | 84.33 (22.591)
  Female: Year 6: number analyzed (Participants) | 2
  Female: Year 6 | 106.00 (22.627)
  Female: Year 7: number analyzed (Participants) | 2
  Female: Year 7 | 77.50 (19.092)
  Female: Year 8: number analyzed (Participants) | 1
  Female: Year 8 | 73.70 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Female: Year 8.5: number analyzed (Participants) | 0

14. Secondary Outcome: C-terminal Telopeptide (CTX) Values of Recombinant Human Growth Hormone (r-hGH) Treated Subjects With Hypochondroplasia (HCH) From Year 1 up to 9.5 Years
Description: CTX (Blood) as bone marker was analyzed with the Immunology system Elecsys. Data was reported by gender. Male subjects were analyzed till 9.5 years and female subjects were analyzed till 8.5 years.
Time Frame: Year 1, 2, 3, 4, 5, 6, 7, 8 (both male and female); 8.5 (only for female), 9 (only for male), 9.5 (only for male)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: picomole per liter (pmol/L)
Arm/Group | r-hGH (Saizen®)
Number analyzed (Participants) | 19
picomole per liter (pmol/L)
  Male: Year 1: number analyzed (Participants) | 6
  Male: Year 1 | 15784.17 (1426.214)
  Male: Year 2: number analyzed (Participants) | 8
  Male: Year 2 | 16304.13 (2537.725)
  Male: Year 3: number analyzed (Participants) | 8
  Male: Year 3 | 15703.50 (3249.336)
  Male: Year 4: number analyzed (Participants) | 4
  Male: Year 4 | 15868.25 (4485.621)
  Male: Year 5: number analyzed (Participants) | 4
  Male: Year 5 | 17088.75 (5208.676)
  Male: Year 6: number analyzed (Participants) | 2
  Male: Year 6 | 12361.00 (4000.810)
  Male: Year 7: number analyzed (Participants) | 1
  Male: Year 7 | 13795.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Male: Year 8: number analyzed (Participants) | 1
  Male: Year 8 | 15345.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Male: Year 9: number analyzed (Participants) | 1
  Male: Year 9 | 15655.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Male: Year 9.5: number analyzed (Participants) | 1
  Male: Year 9.5 | 17205.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Female: Year 1: number analyzed (Participants) | 9
  Female: Year 1 | 16008.00 (2725.874)
  Female: Year 2: number analyzed (Participants) | 11
  Female: Year 2 | 15183.09 (4371.058)
  Female: Year 3: number analyzed (Participants) | 11
  Female: Year 3 | 12595.18 (3172.529)
  Female: Year 4: number analyzed (Participants) | 4
  Female: Year 4 | 13911.00 (1076.509)
  Female: Year 5: number analyzed (Participants) | 3
  Female: Year 5 | 12503.33 (2867.849)
  Female: Year 6: number analyzed (Participants) | 2
  Female: Year 6 | 13678.50 (603.162)
  Female: Year 7: number analyzed (Participants) | 2
  Female: Year 7 | 13446.50 (931.260)
  Female: Year 8: number analyzed (Participants) | 1
  Female: Year 8 | 11858.00 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed at the specified time point.
  Female: Year 8.5: number analyzed (Participants) | 0

15. Secondary Outcome: Number of Subjects With Fibroblast Growth Factor Receptor (FGFR3) Mutation
Description: Genetic analysis was performed to record FGFR3 gene mutation. Genomic DNA was extracted from lymphocytes of collected blood samples using standard procedures. A set of intronic primers was designed based on the genomic sequence of the human FGFR3 gene and used to amplify exons 2-19. Number of subjects with FGFR3 mutation were reported.
Time Frame: Baseline up to 3 years
Population: as for baseline characteristics
Measure: Number; unit: Subjects
Arm/Group | r-hGH (Saizen®)
Number analyzed (Participants) | 19
Subjects | 14

16. Secondary Outcome: Number of Subjects With Adverse Event (AE) and Serious Adverse Event (SAE)
Description: AEs: any new untoward medical occurrences/worsening of pre-existing medical condition, whether or not related to study drug , SAE: any AE that resulted in death; was life threatening; resulted in persistent/significant disability/incapacity; resulted in/prolonged an existing in-patient hospitalization; was a congenital anomaly/birth defect; or was an overdose.
Time Frame: Baseline up to 9.5 years
Population: as for baseline characteristics
Measure: Number; unit: Subjects
Arm/Group | r-hGH (Saizen®)
Number analyzed (Participants) | 19
Subjects
  AEs | 18
  SAEs | 1

ADVERSE EVENTS:
Arm/Group | r-hGH (Saizen®)
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 1/19
Other Adverse Events (participants affected / at risk) | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | r-hGH (Saizen®) (N=19)
Abdominal pain (Gastrointestinal disorders) | 1
Appendicitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | r-hGH (Saizen®) (N=19)
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombopenia (Blood and lymphatic system disorders) | 1
Leucopenia (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Precocious puberty (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Dental cyst (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 3
Fatigue (General disorders) | 1
Oedema peripheral (General disorders) | 1
Tooth abscess (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Vulvitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 3
Gastroenteritis (Infections and infestations) | 3
Rhinitis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 2
Meningitis viral (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Appendicitis (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1
Insulin-like growth factor increased (Investigations) | 3
Vitamin D deficiency (Metabolism and nutrition disorders) | 3
Insulin resistance (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Foot deformity (Musculoskeletal and connective tissue disorders) | 1
Knee deformity (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Torticollis (Musculoskeletal and connective tissue disorders) | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 5
Limb deformity (Metabolism and nutrition disorders) | 1
Deformity thorax (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Lordosis (Musculoskeletal and connective tissue disorders) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 4
Sciatica (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Anger (Psychiatric disorders) | 1
Gynaecomastia (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Corrective lens user (Social circumstances) | 1
Mole excision (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other